CLINICAL TRIAL: NCT01666860
Title: Long-term Follow-up of the Anterior Lumbar Interbody Fusion Procedure.
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/740
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Anterior Lumbar Interbody Fusion Procedure
Keywords: anterior lumbar interbody fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anterior Lumbar Interbody Fusion procedure
  Interventions: Procedure: Anterior Lumbar Interbody Fusion procedure

INTERVENTIONS:
Procedure: Anterior Lumbar Interbody Fusion procedure

SUMMARY:
During the period 1989-1999, a number of patients underwent an ALIF-procedure. Anterior Lumbar Interbody Fusion procedure (ALIF) is a type of lumbar spinal fusion. The approach of the lumbar region is by incision of the abdominal wall. The intervertebral disc is removed and replaced by a bone graft. These patients form the population of this study. The goal of this study is to evaluate their current medical condition and to determine the clinical outcome.

The clinical result will be stipulated by means of standardized questionnaires (VAS-score, Oswestry low Back Pain Questionnaire and SF-36)

ELIGIBILITY:
Inclusion Criteria:

* An Anterior Lumbar Interbody Fusion procedure between 1999 and 2005

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have an Anterior Lumbar Interbody Fusion Procedure as treatment for degenerative disc disease.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
A clinical evaluation before an Anterior Lumbar Interbody Fusion procedure. | Baseline
  The clinical result will be stipulated by means of standardized questionnaires.
A clinical evaluation after an Anterior Lumbar Interbody Fusion procedure. | 5 years after the operation
  The clinical result will be stipulated by means of standardized questionnaires.

SECONDARY OUTCOMES:
Union of the vertebrae. | 1 day (At the standard follow up consultation)
  Standard post operative X-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Poffyn, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be